CLINICAL TRIAL: NCT04120090
Title: Clinical Study of Different Doses of Ruxolitinib as a Salvage Therapy for Refractory/Relapsed Hemophagocytic Lymphohistiocytosis
Brief Title: Ruxolitinib as a Salvage Therapy for Hemophagocytic Lymphohistiocytosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Clinical Professor, Beijing Friendship Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ruxolitinib-HLH
Record Dates: First submitted 2019-10-06; First posted 2019-10-09 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Hemophagocytic Lymphohistiocytosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose (Active Comparator)
  Interventions: Drug: low dose ruxolitinib
- High dose (Experimental)
  Interventions: Drug: high dose ruxolitinib

INTERVENTIONS:
Drug: low dose ruxolitinib — The dose for adult patients(Age>=14 years) is generally 10 mg twice daily. For children(Age<14 years ,weight >=25kg),the dose was generally 5mg twice daily. For children(Age<14 years, weight <25kg), the dose was generally 2.5mg twice daily.
  Arms: Low dose
Drug: high dose ruxolitinib — The dose for adult patients(Age>=14 years) is generally 20mg twice daily. For children(Age<14 years ,weight >=25kg),the dose was generally 10mg twice daily. For children(Age<14 years, weight <25kg), the dose was generally 5mg twice daily
  Arms: High dose

SUMMARY:
This study aimed to investigate the efficacy and safety of different doses of ruxolitinib as a salvage therapy for refractory/relapsed hemophagocytic lymphohistiocytosis(HLH).

ELIGIBILITY:
Inclusion Criteria:

1. meet hemophagocytic lymphohistiocytosis (HLH)-04 diagnostic criteria;
2. treated with HLH-94 no less than 2 weeks before enrollment and did not achieve at least PR; or relapsed patients after remission；
3. Life expectancy exceeds 1 month;
4. Age≥1 year old and ≤75 years old, gender is not limited；
5. Before the start of the study, total bilirubin ≤ 10 times the upper limit of normal; serum creatinine ≤ 1.5 times normal；
6. Serum human immunodeficiency virus(HIV) antigen or antibody negative；
7. Hepatitis C virus (HCV) antibody is negative, or HCV antibody is positive, but HCV RNA is negative；
8. Both hepatitis B virus (HBV) surface antigen and HBV core antibody were negative. If any of the above is positive, peripheral blood hepatitis B virus DNA titer should be detected, and less than 1×103 copies/ml can enter the group；
9. Informed consent.

Exclusion Criteria:

1. Pregnancy or lactating Women；
2. Allergic to ruxolitinib；
3. Active bleeding of the internal organs；
4. uncontrollable infection；
5. Serious mental illness;
6. Non-melanoma skin cancer history;
7. Patients unable to comply during the trial and/or follow-up phase;
8. Participate in other clinical research at the same time.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | 1 years
  complete response (CR) and partial response (PR) rates
Progression Free Survival | 1 years
  from date of inclusion to date of progression, relapse, or death from any cause Overall Survival

SECONDARY OUTCOMES:
Overall Survival | 1 years
  from the date of inclusion to date of death, irrespective of cause Adverse Events
Adverse events | 1 year
  Adverse events including myelosuppression, infection, bleeding and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No